CLINICAL TRIAL: NCT02317276
Title: A Study in Atopic Dermatitis to Determine Serum and Skin Biopsy Biomarkers in Patients Receiving Topical Corticosteroid (TCS) and Following TCS Withdrawal
Brief Title: A Study to Determine Serum and Skin Biopsy Biomarkers in Patients Receiving Topical Corticosteroid (TCS) and Following TCS Withdrawal
Acronym: GNE-AD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to meet the study's recruitment goals
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GNE AD 431
Record Dates: First submitted 2014-12-03; First posted 2014-12-15 (Estimated); Results first posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Triamcinolone; Ointments

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Topical Triamcinolone 0.1% ointment will be provided for twice daily application, during treatment periods.
  Interventions: Drug: Triamcinolone 0.1%

INTERVENTIONS:
Drug: Triamcinolone 0.1% — Topical ointment
  Other Names: Triamcinolone 0.1% ointment

SUMMARY:
The purpose of this study is to assess the differential expression of AD biomarkers in serum, plasma, and skin biopsies from both lesional and non-lesional skin in moderate to severe AD patients in the presence of TCS and after withdrawal from TCS.

DETAILED DESCRIPTION:
This exploratory study consists of four visits to the investigator site post screening: at Weeks 0 (baseline), 2, 6 and 8 (Figure 1). At the first visit (baseline), patients who have met the screening eligibility criteria will be started on a stable TCS regimen for a total of two weeks. At the second visit (Week 2) following two weeks of therapy on stable TCS, patients will stop TCS and blood, serum, plasma and two 6mm punch biopsies (one lesional (L) and one non-lesional (NL) skin) will be obtained. At the third visit (Week 6), after four weeks receiving no TCS, the same sample collections will be repeated and the patients will then enter a two week safety follow up. At the end of the safety follow up (last visit, Week 8) and after obtaining written informed consent by the patient, blood, serum and plasma samples mav be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18-75 years of age
2. AD diagnosed by the Rajka/Hanifin criteria at the time of screening and that has been present for at least 1 year
3. History of inadequate response to a stable regimen of TCS for 1 month (in the 3 months immediately preceding the screening visit) as treatment for their AD
4. Eczema Area and Severity Index (EASI) score ≥ 14 at the screening and baseline visits
5. Investigator's Global Assessment (IGA; 5-point) score ≥ 3 at the screening and baseline visits
6. ≥10% body surface area involvement by AD
7. A washout period prior to screening for those patients who have previously received the following medications:

   * Cyclosporine/Oral Steroids/Imuran/Mycophenolate Mofetil/Other systemic immunosuppressants: 4 weeks
   * Phototherapy: 4 weeks
   * Biologics: 5 half lives of the drug

Exclusion Criteria:

1. Evidence of other concomitant skin conditions (e.g., psoriasis or contact dermatitis)
2. Use of topical calcineurin inhibitors within 4 weeks of screening
3. Hypersensitivity to TCS or to any other ingredients contained by the emollient or TCS product used during the study
4. Evidence of active skin infection at screening or baseline visit
5. Evidence or history of active or latent infections such as tuberculosis or hepatitis C
6. Patient clinical condition is not appropriate for treatment with protocol prescribed TCS
7. Use of an investigational agent within 4 weeks prior to screening or within 5 half-lives of the investigational agent, whichever is longer
8. Use of a tanning booth/parlor within 4 weeks before the baseline visit
9. Use of any anti-histamine medication within 4 weeks before the baseline visit.
10. History of any condition (e.g. bleeding diathesis) that may predispose the patient to complications associated with the planned skin biopsy procedures
11. Known current malignancy or current evaluation for a potential malignancy, including basal or squamous cell carcinoma of the skin or carcinoma in situ
12. Other clinically significant medical disease that is uncontrolled despite treatment that is likely, in the opinion of the investigator, to impact the patient's ability to participate in the study or to impact the study pharmacodynamic (PD), or safety assessments
13. Unwillingness or inability to comply with the study protocol for any other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-12; Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Arron, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Dermatology, San Francisco, California, United States

REFERENCES:
- [Result] Bieber T. Atopic dermatitis. N Engl J Med. 2008 Apr 3;358(14):1483-94. doi: 10.1056/NEJMra074081. No abstract available. PMID 18385500
- [Result] Williams DL, Ozment-Skelton T, Li C. Modulation of the phosphoinositide 3-kinase signaling pathway alters host response to sepsis, inflammation, and ischemia/reperfusion injury. Shock. 2006 May;25(5):432-9. doi: 10.1097/01.shk.0000209542.76305.55. PMID 16680006
- [Result] Simpson EL. Atopic dermatitis: a review of topical treatment options. Curr Med Res Opin. 2010 Mar;26(3):633-40. doi: 10.1185/03007990903512156. PMID 20070141
- [Result] Ring J, Alomar A, Bieber T, Deleuran M, Fink-Wagner A, Gelmetti C, Gieler U, Lipozencic J, Luger T, Oranje AP, Schafer T, Schwennesen T, Seidenari S, Simon D, Stander S, Stingl G, Szalai S, Szepietowski JC, Taieb A, Werfel T, Wollenberg A, Darsow U; European Dermatology Forum (EDF); European Academy of Dermatology and Venereology (EADV); European Federation of Allergy (EFA); European Task Force on Atopic Dermatitis (ETFAD); European Society of Pediatric Dermatology (ESPD); Global Allergy and Asthma European Network (GA2LEN). Guidelines for treatment of atopic eczema (atopic dermatitis) part I. J Eur Acad Dermatol Venereol. 2012 Aug;26(8):1045-60. doi: 10.1111/j.1468-3083.2012.04635.x. PMID 22805051
- [Result] Schneider L, Tilles S, Lio P, Boguniewicz M, Beck L, LeBovidge J, Novak N, Bernstein D, Blessing-Moore J, Khan D, Lang D, Nicklas R, Oppenheimer J, Portnoy J, Randolph C, Schuller D, Spector S, Tilles S, Wallace D. Atopic dermatitis: a practice parameter update 2012. J Allergy Clin Immunol. 2013 Feb;131(2):295-9.e1-27. doi: 10.1016/j.jaci.2012.12.672. PMID 23374261
- [Result] Gittler JK, Shemer A, Suarez-Farinas M, Fuentes-Duculan J, Gulewicz KJ, Wang CQ, Mitsui H, Cardinale I, de Guzman Strong C, Krueger JG, Guttman-Yassky E. Progressive activation of T(H)2/T(H)22 cytokines and selective epidermal proteins characterizes acute and chronic atopic dermatitis. J Allergy Clin Immunol. 2012 Dec;130(6):1344-54. doi: 10.1016/j.jaci.2012.07.012. Epub 2012 Aug 27. PMID 22951056
- [Result] Choy DF, Hsu DK, Seshasayee D, Fung MA, Modrusan Z, Martin F, Liu FT, Arron JR. Comparative transcriptomic analyses of atopic dermatitis and psoriasis reveal shared neutrophilic inflammation. J Allergy Clin Immunol. 2012 Dec;130(6):1335-43.e5. doi: 10.1016/j.jaci.2012.06.044. Epub 2012 Aug 22. PMID 22920495

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For this study we recruited participants from UCSF Dermatology Clinic, and by posting advertisements online
Pre-assignment Details: There was a washout period prior to screening for those patients who have previously received the following medications:
  1. Cyclosporine/Oral Steroids/Imuran/Mycophenolate Mofetil/Other systemic immunosuppressants: 4 weeks
  2. Phototherapy: 4 weeks
  3. Biologics: 5 half lives of the drug
Period: Overall Study
Arm/Group | Treatment
Started | 11
Completed | 5
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Eczema Area and Severity Index (EASI) [Mean (Standard Deviation); unit: scores on a scale] — The EASI score measures extent of eczema involvement and severity of eczema signs, per body region. The body regions are head/neck, trunk, upper extremities, and lower extremities. Area of eczema involvement is scored as a % where 1= 1-9% involvement, 2= 10-29%, 3= 30-49%, 4= 50-69%, 5= 70-89%, 6= 90-100%. Severity of eczema signs is scored as number 0-3 where 0=none, 1=mild, 2=moderate, 3=severe. The % and severity are then added and multiplied with a multiplier for a total score. The total score ranges from 0-72. A higher score indicates more involved and more severe eczema, a worse outcome.
  scores on a scale | 19.7 (6.7)
Investigator's Global Assessment (IGA) [Mean (Standard Deviation); unit: scores on a scale] — The Investigator's Global Assessment (IGA) is a 5-point scale measuring disease severity (in this case, eczema severity). A score of 0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe. The number given is the score (not added or multiplied, and half points/scores cannot be used). A higher score indicates more severe eczema and a worse outcome.
  scores on a scale | 3.1 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood and Tissue Levels of Biomarkers Following Treatment of Atopic Dermatitis With Topical Corticosteroids.
Description: The blood and skin biomarkers to be evaluated include but are not limited to eosinophils, Immunoglobulin E (IgE), Interleukin 13 (IL-13), Chemokine ligand 13 (CCL-13), and Chemokine ligand 17 (CCL-17). These biomarkers will be evaluated for differential gene expression and protein levels in samples obtained from atopic dermatitis patients on and off topical corticosteroid treatment.
Time Frame: Baseline to Week 8
Population: No samples were analyzed for the primary outcome measure of change in blood and tissue levels. Since the study was terminated, the blood and tissue samples were not analyzed as planned.
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 1 year, during the duration of the study.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

LIMITATIONS AND CAVEATS:
Due to our inability to meet the sponsor's recruitment goals, the study was terminated and no data was analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-05): https://cdn.clinicaltrials.gov/large-docs/76/NCT02317276/Prot_SAP_000.pdf